CLINICAL TRIAL: NCT05158426
Title: Application of the Propofol Precise Infusion Model
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Du, professor, West China Hospital
Other Study IDs: WestChinaH-2018-1
Record Dates: First submitted 2021-11-18; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Propofol Overdose of Undetermined Intent
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sample
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- propofol susceptibility group: patients undergoing gastrointestinal endoscopy
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — anesthesia induction is initiated with intravenous infusion propofol at 1.5µg/ml, and increased 0.5µg/ml every 3min until OAA/S score 0.
  Other Names: Diprivan

SUMMARY:
Propofol is one of the most commonly used anesthetics in the world. However, the dose-response of propofol was remarkable variety. Herein, this study aims to investigate the possible association of gene polymorphism and propofol susceptibility, and to research more precise infusion model of this drug.

DETAILED DESCRIPTION:
Patients undergoing gastrointestinal endoscopy will be recruited. Anesthesia is induced with propofol via TCI at 1.5µg/ml, and increases 0.5µg/ml for every 3min until OAA/S score 0. During this period, OAA/S score will be evaluated every 1min until OAA/S score 0. At this moment, the blood concentration of propofol, the doses of propofol, the onset time and BIS are recorded, and blood sample for gene polymorphism detection were required.

ELIGIBILITY:
Inclusion Criteria:

1. patients who undergoing gastrointestinal endoscopy with anesthesia
2. age ≥18 years

Exclusion Criteria:

1. hepatic or kidney function injured;
2. received hypnotic sedative drug regularly;
3. Pregnancy, excessive drinking, or current smoker;
4. be allergic to propofol
5. patients who with difficulty communication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who will undergo gastrointestinal endoscopy with propofol
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
gene polymorphism of propofol susceptibility | from anesthesia induction to the end of the gastrointestinal endoscopy
  combination of the blood concentration of propofol (ng/ml) with the onset time(min) at OAA/S score of 0 to demonstrate propofol susceptibility, the gene polymorphism of propofol susceptibility will be detected with the blood sample of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Li, Study Director — West China Hospital; lin Zhang, Study Director — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China